CLINICAL TRIAL: NCT01067274
Title: A Randomized Multicenter Phase III Study to Evaluate the Role of All-trans Retinoic Acid (ATRA) in Combination With Induction Chemotherapy, or Azacitidine and Idarubicin as Salvage Therapy and Idarubicin With Cytarabine or Azacitidine as Maintenance Therapy in Older Patients With Acute Myeloblastic Leukemia (AML)
Brief Title: ALFA-0703 Study in Older Patients With Acute Myeloblastic Leukemia (AML)
Acronym: ALFA-0703
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study abandoned
Sponsor: Acute Leukemia French Association (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Dr Claude GARDIN, Avicenne Hospital- Hôpital Avicenne, AP-HP Bobigny
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALFA-0703 Study - P060205
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2010-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Aged of 65 to 79 years; Older Patients with Acute Myeloblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Tretinoin; Azacitidine; Cytarabine

ARMS (6):
- R1 Arm A : ATRA (Experimental): Idarubicin: 9 mg/m2/d D1 to D4 Cytarabine : 200 mg/m2/d Continuous IV from D1 to D7 Peg-filgrastim : 6 mg SC D9 or filgrastim 5ug/kg/d SC or lenograstim 263ug/d IV 30mn, both from D9 to myeloid recovery(PMN >1G/l over 2 days at minimum
  All-trans retinoic acid (ATRA): 45mg/m2/day in two divided doses from D8 to D28
  Interventions: Drug: Vesanoid (ATRA)
- R1 Arm B : no ATRA (No Intervention): Idarubicin: 9 mg/m2/d D1 to D4 Cytarabine : 200 mg/m2/d Continuous IV from D1 to D7 Peg-filgrastim : 6 mg SC D9 or filgrastim 5ug/kg/d SC or lenograstim 263ug/d IV 30mn, both from D9 to myeloid recovery(PMN >1G/l over 2 days at minimum
- R2 Arm 1A : AZACITIDINE and ATRA (Experimental): Azacitidine: 75 mg/m2/12h SC from D1 to D5 Idarubicine: 9 mg/m2/d IV on D5 All-trans retinoic acid (ATRA): 45mg/m2/d in two divided doses from D8 to D21
  Interventions: Drug: Vesanoid (ATRA); Drug: AZACITIDINE (VIDAZA)
- R2 Arm 1B : AZACITIDINE and No ATRA (Experimental): Azacitidine: 75 mg/m2/12h SC from D1 to D5 Idarubicine: 9 mg/m2/d IV on D5
  Interventions: Drug: AZACITIDINE (VIDAZA)
- R2 Arm 2A : ATRA (Experimental): Idarubicine : 9 mg/m2/d IV on D1 Cytarabine : 60 mg/m2/12h SC from D1 to D5 All-trans retinoic acid (ATRA): 45mg/ m2/d in two divided doses from D8 to D21
  Interventions: Drug: Vesanoid (ATRA); Drug: CYTARABINE
- R2 Arm 2B : no ATRA (Experimental): Idarubicine : 9 mg/m2/d IV on D1 Cytarabine : 60 mg/m2/12h SC from D1 to D5
  Interventions: Drug: CYTARABINE

INTERVENTIONS:
Drug: Vesanoid (ATRA) — 45 mg/m2/day in two divided doses from D8 to D28
  Other Names: VEZANOIDE
  Arms: R1 Arm A : ATRA; R2 Arm 1A : AZACITIDINE and ATRA; R2 Arm 2A : ATRA
Drug: AZACITIDINE (VIDAZA) — 75 mg/m2/12h SC from D1 to D5
  Arms: R2 Arm 1A : AZACITIDINE and ATRA; R2 Arm 1B : AZACITIDINE and No ATRA
Drug: CYTARABINE — Cytarabine : 60 mg/m2/12h SC from D1 to D5
  Arms: R2 Arm 2A : ATRA; R2 Arm 2B : no ATRA

SUMMARY:
A Randomized Multicenter Phase III Study to Evaluate the Role of All-trans Retinoic Acid (ATRA) in Combination with Induction Chemotherapy, or Azacitidine and Idarubicin as salvage therapy and Idarubicin with Cytarabine or Azacitidine as Maintenance Therapy in Older Patients with Acute Myeloblastic Leukemia (AML).

To compare the outcome of elderly patients with newly-diagnosed AML treated with standard induction chemotherapy and post-remission therapy, in only patients in CR, with either azacitidine or cytarabine combined to idarubicin +/- ATRA and salvage therapy with azacitidine combined to idarubicin +/- ATRA.

DETAILED DESCRIPTION:
Induction therapy :

First randomization (R1) at baseline : ATRA versus no ATRA.

Salvage therapy :

No conventional salvage therapy is planned. Patients who will not achieve CR, according to IWG criteria after induction will be treated with 3 courses of azacitidine and idarubicin +/- ATRA combination, if eligible for further treatment.

Followed by 3 identical courses and 6 courses of maintenance by azacitidine alone to be delivered every 28 days, in those patients reaching CR or PR after 3 courses (evaluation of response from 28 to 56 days from course 3).

Randomization R2: type of maintenance:

Response to induction will be evaluated 2 weeks after myeloid recovery, just before first consolidation course, due use of to pegfilgrastim, lenograstim or filgrastim during induction.

Responses will be classified according to the Revised Recommendations of the IWG for AML.

Patients in CR only will be subjected to a second randomization R2 as follows 6 courses of combined chemotherapy, will be delivered as outpatients, ATRA according to R1 randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Aged of 65 to 79 years
2. With a morphologically proven diagnosis of AML according to WHO classification either de novo or AML with "myelodysplasia related changes"
3. Not previously treated for AML
4. Signed informed consent.

Exclusion Criteria:

1. APL in the WHO classification.
2. Ph1-positive AML or prior Ph1-positive disease
3. AML evolving from a prior MPN in the WHO 2008 classification.
4. Prior treatment with chemotherapy or radiotherapy for another tumor
5. Prior tumor, if not stable for at least two years, except in-situ carcinoma and skin carcinoma
6. Prior advanced malignant hepatic tumor
7. ECOG Performance Status Score > 2
8. Creatinine level more than 2x's the upper limit of the normal range (ULN) at the laboratory where the analysis was performed, except if AML-related.
9. Total serum bilirubin more than 2x's the ULN at the laboratory where the analysis was performed, except if AML-related.
10. AST (SGOT) or ALT (SGPT) more than 2.5x's the ULN at the laboratory where the analysis was performed, except if AML-related
11. LVEF less than.55 or equivalent by doppler echocardiography
12. Known intolerance to Azacitidine, mannitol, retinoids
13. Positive serum test for HIV and HTLV-1
14. NYHA Grade 3/4 cardiac disease .
15. Severe infection at inclusion time.
16. Psychiatric disease or an history of non-compliance to medical regimens or patients considered potentially unreliable.
17. Absence of health care insurance (affiliation à un régime de Sécurité Sociale)
18. Participation to any study requiring informed consent

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
For randomization R1, the primary endpoint is Event-free Survival (EFS) | 2-year EFS
For randomization R2, the primary endpoint is disease free survival (DFS) | 2-year DFS

SECONDARY OUTCOMES:
Complete Response (CR) rate | 2 years
Overall survival | 2 years
Response rate to azacitidine idarubicin +/-ATRA combination after intensive chemotherapy failure and identification of possible predictors of response to this therapy | 2 years
Assess the safety of combination ATRA + chemotherapy or idarubicin-azacitidine courses and of maintenance with azacitidine | 2 years
Effects on relapse rates of ATRA and maintenance, with respect to cytogenetics risk groups, subtypes of AML and mutational status (FLT3, MLL), and biomarkers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GARDIN CLAUDE, MD, Principal Investigator — Acute Leukemia French Association
Locations (26):
- France (26):
  - Chu Amiens Sud, Amiens
  - CH, Argenteuil
  - Hopital Avicenne, Bobigny
  - Chu Boulogne Sur Mer, Boulogne-sur-Mer
  - CH, Caen
  - Hopital Percy, Clamart
  - Ch Sud Francilien, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - Ch Dunkerque, Dunkirk
  - CH, Lens
  - CHU, Lille
  - CH, Limoges
  - Hopital Edouard Herriot, Lyon
  - CH, Meaux
  - Centre Antoine Lacassagne, Nice
  - St Antoine Hospital, Paris
  - Necker Hospital, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Saint-Louis, Paris
  - Ch Rene Dubos, Pontoise
  - CH, Roubaix
  - CHU, Rouen
  - CNLCC, Saint-Cloud
  - CH, Valenciennes
  - CH, Versailles
  - IGR, Villejuif